CLINICAL TRIAL: NCT02497404
Title: Epigenetic Priming With 5-Azacytidine Prior to in Vivo T-cell Depleted Allogeneic Stem Cell Transplantation for Patients With High Risk Myeloid Malignancies in Morphologic Remission
Brief Title: Azacytidine Prior to in Vivo T-cell Depleted Allo Stem Cell Transplant for Patients With Myeloid Malignancies in CR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1306014009
Record Dates: First submitted 2015-02-19; First posted 2015-07-14 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Leukemia, Erythroblastic, Acute; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Erythroblastic, Acute; Myelodysplastic Syndromes | interventions — Azacitidine; fludarabine; fludarabine phosphate; Melphalan; Alemtuzumab; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 5 Azacytidine (Experimental): Patients will be given a five day course of subcutaneous 5-azacytidine, followed by a reduced intensity conditioning regimen of fludarabine and melphalan with or without total body irradiation prior to an allogeneic hematopoietic stem cell transplantation from a related or unrelated HLA matched donor.
  Interventions: Drug: 5-Azacytidine; Drug: Fludarabine; Drug: Melphalan; Drug: Alemtuzumab; Radiation: Total Body Irradiation

INTERVENTIONS:
Drug: 5-Azacytidine — Patients will be given a five day course of subcutaneous 5-azacytidine followed by a reduced intensity conditioning regimen of fludarabine and melphalan with or without total body irradiation prior to an allogeneic hematopoietic stem cell transplantation from a related or unrelated HLA matched donor. 5-Azacytidine 75 mg/m2 subcutaneously daily at the same time on days -11, -10, -9,
  -8 and -7. This will be administered on an outpatient basis if possible.
  Other Names: Vidaza
Drug: Fludarabine — Conditioning regimen: Hospital admission will usually take place on the first day of the conditioning regimen. Fludarabine will be given at 40 mg/m2 intravenously daily at the same time over 30 minutes on days -6,-5,-4,-3.
  Other Names: Fludara
Drug: Melphalan — Conditioning regimen: Hospital admission will usually take place on the first day of the conditioning regimen. Melphalan will be given at 140 mg/m2 IV on day -3.
  Other Names: Alkeran
Drug: Alemtuzumab — Conditioning regimen: Hospital admission will usually take place on the first day of the conditioning regimen. Alemtuzumab will be given at 30 mg subcutaneously on Days -4 and -2 for unrelated donors, and Day -2 for related donors.
  Other Names: Campath, Lemtrada
Radiation: Total Body Irradiation — Conditioning regimen: Hospital admission will usually take place on the first day of the conditioning regimen. Total Body Irradiation (TBI) will be given at 2 doses of 200 cGy each on one day of the conditioning regimen (between days -6 and -3).
  Other Names: TBI

SUMMARY:
The purpose of this study is to determine whether 5-Azacytidine priming before the conditioning regimen for subjects receiving a hematopoietic stem cell transplant is an effective treatment for high risk myeloid malignancies in complete remission (CR).

DETAILED DESCRIPTION:
This open label two-step phase II study is designed to determine the safety and efficacy of epigenetic priming with 5-Azacytidine immediately prior to reduced intensity conditioning for an in vivo T-cell depleted hematopoietic stem cell transplantation for high risk myeloid malignancies in complete remission (CR).

Subjects will be given a five day course of subcutaneous 5-azacytidine, followed by a reduced intensity conditioning regimen of fludarabine, melphalan and total body irradiation (TBI) prior to an allogeneic hematopoietic stem cell transplantation from a related or unrelated Human Leukocyte Antigen (HLA) matched donor.

The effect of 5-azacytidine on global gene methylation will be assessed. Evaluations for safety, in particular for graft failure, transplant related mortality and acute graft versus host disease will be made on a weekly basis. Efficacy, as defined by disease free survival, will be evaluated with a bone marrow biopsy at the standard time points, which are one-, three-, six-, and twelve-months after transplant and upon clinical suspicion within regular follow-up visits - weekly for the first 3 months, then biweekly for 3 months, then monthly until one-year post-stem cell transplant. Thereafter, unless otherwise dictated by the clinical scenario, the follow up visits will be every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) as specified below:

  1. Acute myeloid leukemia with poor risk cytogenetics in complete morphologic remission. These include: del (5q)/-5, del (7q)/-7, abn 3q, 9q, 11q, 20q, 21q, 17p, t(6;9), t(9;22) or complex karyotypes (≥ 3 unrelated abnormalities); or
  2. Acute myeloid leukemia with either Flt-3, TET-2, p53, DNMT3A, or ASXL1 mutation, mutations of genes involved in the chromatin/spliceosome category (EZH2, SRSF2, U2AF1, ZRSR2), BCOR, and RUNX1, as well as MLL rearrangement, EVI1 overexpression in complete morphologic remission; or
  3. Acute myeloid leukemia with a white blood cell count of greater than or equal to 50,000/mcL at presentation in first complete morphologic remission; or
  4. Acute myeloid leukemia in first complete morphologic remission, having required more than one course of induction chemotherapy to attain remission status; or
  5. Acute myeloid leukemia, all types, excluding M3 (Promyelocytic leukemia) in second or higher complete morphologic remission; or
  6. Myelodysplastic syndromes (intermediate-2, high risk and chronic myelomonocytic leukemia (CMML) with bone marrow blasts <5%); or
  7. Secondary acute myeloid leukemia on the basis of prior MDS or prior myeloproliferative neoplasm (MPN) in complete morphologic remission
* Life expectancy not severely limited by concomitant disease
* Karnofsky Performance Score greater than or equal to 70%.
* Adequate organ function as defined below:

Serum Bilirubin:<2.0 mg/dL; Alanine Aminotransferase (ALT) (SGPT): <3 x upper limit of normal; Creatinine Clearance:>60 mL/min (eGFR as estimated by the modified Modification of Diet in Renal Disease Study (MDRD) equation)

- Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Evidence of chronic active hepatitis or cirrhosis
* HIV infection
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and lactating women are excluded from the study because the risks to an unborn fetus or potential risks in nursing infants are unknown.
* There are no prior therapies or concomitant medications that would render the patients ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02-13 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2021-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Mayer, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 Azacytidine: Patients will be given a five day course of subcutaneous 5-azacytidine, followed by a reduced intensity conditioning regimen of fludarabine and melphalan with or without total body irradiation (TBI) prior to an allogeneic hematopoietic stem cell transplantation from a related or unrelated HLA matched donor.
  5-Azacytidine: Patients will be given a five day course of subcutaneous 5-Azacytidine followed by a reduced intensity conditioning regimen of fludarabine and melphalan with or without total body irradiation prior to an allogeneic hematopoietic stem cell transplantation from a related or unrelated HLA matched donor. AZA 75 mg/m2 subcutaneously daily at the same time on days -11, -10, -9, -8 and -7. This will be administered on an outpatient basis if possible.
  Fludarabine (conditioning regimen): Fludarabine will be given at 40 mg/m2 intravenously daily at the same time over 30 minutes on days -6,-5,-4,-3.
  Melphalan (conditioning regimen): Melphalan will be given at 140 mg/m2 IV on day -3.
  Alemtuzumab (conditioning regimen): Alemtuzumab will be given at 30 mg subcutaneously on Days -4 and -2 for unrelated donors, and Day -2 for related donors.
  TBI (conditioning regimen): TBI will be given at 2 doses of 200 cGy each on one day of the conditioning regimen (between days -6 and -3).
Period: Overall Study
Arm/Group | 5 Azacytidine
Started | 40
Completed | 39
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | 5 Azacytidine
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 35
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40
Disease [Count of Participants; unit: Participants] — Hematologic malignancy that allogeneic hematopoietic stem cell transplant is intended to treat
  Participants
    Acute Myeloid Leukemia | 34
    Myelodysplastic Syndrome/Myeloproliferative Disease | 6
Donor Relationship [Count of Participants; unit: Participants] — Donor relationship to participant for allogeneic stem cell transplant Population: One participant was removed from the study before stem cell transplantation and is therefore unevaluable for this baseline measure
  Participants
    number analyzed (Participants) | 39
    Matched Related Donor | 17
    Matched Unrelated Donor | 22

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival at 1 Year Post-transplant
Description: Number of participants without evidence of progression of underlying malignancy for which the transplant was performed, assessed at 1 year post-transplant.
Time Frame: 1 year post-transplant
Population: 1 participant was unevaluable as they were removed from study before undergoing hematopoietic stem cell transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Azacytidine
Number analyzed (Participants) | 39
Participants | 18
Statistical Analysis 1: Comparison: 5 Azacytidine; Test type: Other — Clopper-Pearson (exact) 95% confidence interval provided for the survival proportion; Proportion (percent) = 46.2, 95% CI 2-sided [30.1 to 62.8]

2. Secondary Outcome: Disease Free Survival at 6 Months Post-transplant
Description: Number of participants without evidence of progression of underlying malignancy for which the transplant was performed, assessed at 6 months post-transplant
Time Frame: 6 months post-transplant
Population: 1 participant was unevaluable as they were removed from study before undergoing hematopoietic stem cell transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Azacytidine
Number analyzed (Participants) | 39
Participants | 25
Statistical Analysis 1: Comparison: 5 Azacytidine; Test type: Other — Clopper-Pearson (exact) 95% confidence interval provided for the survival proportion; Proportion (percent) = 64.1, 95% CI 2-sided [47.2 to 78.8]

3. Secondary Outcome: Disease Free Survival at 2 Years Post-transplant
Description: Number of participants without evidence of progression of underlying malignancy for which the transplant was performed, assessed at 2 years post-transplant.
Time Frame: 2 years post-transplant
Population: 1 participant was unevaluable as they were removed from study before undergoing hematopoietic stem cell transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Azacytidine
Number analyzed (Participants) | 39
Participants | 13
Statistical Analysis 1: Comparison: 5 Azacytidine; Test type: Other — Clopper-Pearson (exact) 95% confidence interval provided for the survival proportion; Proportion (percent) = 33.3, 95% CI 2-sided [19.1 to 50.2]

4. Secondary Outcome: Overall Survival at 6 Months Post-transplant
Description: Number of participants alive at 6 months post-transplant
Time Frame: 6 months post-transplant
Population: 1 participant was unevaluable as they were removed from study before undergoing hematopoietic stem cell transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Azacytidine
Number analyzed (Participants) | 39
Participants | 35
Statistical Analysis 1: Comparison: 5 Azacytidine; Test type: Other — Clopper-Pearson (exact) 95% confidence interval provided for the survival proportion; Proportion (percent) = 89.7, 95% CI 2-sided [75.8 to 97.1]

5. Secondary Outcome: Overall Survival at 1 Year Post-Transplant
Description: Number of participants alive at 1 year post-transplant
Time Frame: 1 year post-transplant
Population: 1 participant was unevaluable as they were removed from study before undergoing hematopoietic stem cell transplant
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Azacytidine
Number analyzed (Participants) | 39
Participants | 25
Statistical Analysis 1: Comparison: 5 Azacytidine; Test type: Other — Clopper-Pearson (exact) 95% confidence interval provided for the survival proportion; Proportion (percent) = 64.1, 95% CI 2-sided [47.2 to 78.8]

6. Secondary Outcome: Overall Survival at 2 Years Post-Transplant
Description: Number of participants alive at 2 years post-transplant
Time Frame: 2 years post-transplant
Population: 1 participant was unevaluable as they were removed from study before undergoing hematopoietic stem cell transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Azacytidine
Number analyzed (Participants) | 39
Participants | 15
Statistical Analysis 1: Comparison: 5 Azacytidine; Clopper-Pearson (exact) 95% confidence interval provided for the survival proportion; Test type: Other; Proportion (percent) = 38.5, 95% CI 2-sided [23.4 to 55.4]

7. Secondary Outcome: Graft Failure
Description: Number of patients who experience graft failure, defined as the absence of neutrophil engraftment by Day +21 or a drop in the absolute neutrophil count to <0.3 cells/microL for five consecutive days occurring after initial neutrophil engraftment within the first 3 weeks post-transplantation.
Time Frame: 21 days post-transplant
Population: 1 participant was unevaluable as they were removed from study before undergoing hematopoietic stem cell transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Azacytidine
Number analyzed (Participants) | 39
Participants | 1
Statistical Analysis 1: Comparison: 5 Azacytidine; Test type: Other — Clopper-Pearson (exact) 95% confidence interval provided for the graft failure proportion; Proportion (percent) = 2.6, 95% CI 2-sided [0.07 to 13.5]

8. Secondary Outcome: Acute Graft-versus-Host Disease (GVHD)
Description: Number of patients who develop acute graft-versus-host disease of any grade.
Time Frame: 2 years post-transplant
Population: 1 participant was unevaluable as they were removed from study before undergoing hematopoietic stem cell transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Azacytidine
Number analyzed (Participants) | 39
Participants | 13
Statistical Analysis 1: Comparison: 5 Azacytidine; Test type: Other — Clopper-Pearson (exact) 95% confidence interval provided for the GVHD proportion; Proportion (percent) = 33.3, 95% CI 2-sided [19.1 to 50.2]

9. Secondary Outcome: High-Risk Extensive Chronic Graft-versus-Host-Disease
Description: Number of patients who develop high-risk extensive chronic graft-versus-host disease. Extensive chronic GVHD is defined as generalized skin or multiple organ involvement. High risk chronic GVHD is defined as platelet count of less than 100k/microL
Time Frame: 2 years post-transplant
Population: 1 participant was unevaluable as they were removed from study before undergoing hematopoietic stem cell transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 Azacytidine
Number analyzed (Participants) | 39
Participants | 2
Statistical Analysis 1: Comparison: 5 Azacytidine; Test type: Other — Clopper-Pearson (exact) 95% confidence interval provided for the high-risk extensive chronic graft-versus-host-disease proportion; Proportion (percent) = 5.1, 95% CI 2-sided [0.63 to 15.3]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all patients from start of 5-azacytidine therapy through 5 years post-transplant or when the participant was removed from the study, whichever was sooner.
Description: All adverse events were first documented by the study transplant physicians and thereafter collated and graded by two independent reviewed according to CTCAE version 4.0. Per protocol, events reported were all infectious events and Grade 3 and higher events for non-infectious events
Arm/Group | 5 Azacytidine
All-Cause Mortality (participants affected / at risk) | 28/40
Serious Adverse Events (participants affected / at risk) | 28/40
Other Adverse Events (participants affected / at risk) | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 Azacytidine (N=40)
Atypical Hemolytic Uremic Syndrome (Blood and lymphatic system disorders) | 4 (4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Pericardial Effusion (Cardiac disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Intra-Abdominal Abscess (Gastrointestinal disorders) | 1 (1)
Failure to Thrive (General disorders) | 1 (1)
Hypervolemia (General disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Infusion-Related Reaction (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Bacteremia (Infections and infestations) | 3 (3)
Human Herpesvirus 6 Infection (Infections and infestations) | 1 (1)
Cytomegalovirus Infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3)
Norovirus Infection (Infections and infestations) | 1 (1)
Upper Respiratory Infection - Influenza B (Infections and infestations) | 1 (1)
Upper Respiratory Infection - Rhinovirus (Infections and infestations) | 1 (1)
Fungal Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 5 (5)
Bronchial Infection (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2)
Fungal Infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Herpes Simplex Virus Infection (Infections and infestations) | 1 (1)
Acute Graft-versus-Host Disease (Investigations) | 2 (2)
Platelet Count Decreased (Investigations) | 1 (1)
Chronic Graft-versus-Host Disease (Investigations) | 1 (1)
Post-Transplant Lymphoproliferative Disorder (Investigations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Intracranial Hemorrhage (Nervous system disorders) | 2 (2)
Stroke (Nervous system disorders) | 1 (1)
Posterior Reversible Encephalopathy Syndrome (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 6 (6)
Renal Failure (Renal and urinary disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 Azacytidine (N=40)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Mucositis Oral (Gastrointestinal disorders) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Rectal Pain (Gastrointestinal disorders) | 1 (1)
Periapical Abscess (Gastrointestinal disorders) | 1 (1)
Hepatosplenic Lesion (Hepatobiliary disorders) | 1 (1)
Bacteremia (Infections and infestations) | 11 (11)
Urinary Tract Infection (Infections and infestations) | 7 (7)
Upper Respiratory Infection - Parainfluenza (Infections and infestations) | 8 (8)
Clostridium difficile Colitis (Infections and infestations) | 12 (12)
Adenovirus Infection (Infections and infestations) | 3 (3)
Human Herpesvirus 6 Infection (Infections and infestations) | 13 (13)
Upper Respiratory Infection - Respiratory Synctyial Virus (Infections and infestations) | 3 (3)
Cytomegalovirus Infection (Infections and infestations) | 11 (11)
Varicella Zoster Infection (Infections and infestations) | 1 (1)
Upper Respiratory Infection - Influenza B (Infections and infestations) | 2 (2)
Upper Respiratory Infection - Rhinovirus (Infections and infestations) | 10 (10)
BK Virus Infection (Infections and infestations) | 9 (9)
Upper Respiratory Infection - Human metapneumovirus (Infections and infestations) | 4 (4)
Upper Respiratory Infection - Staphylococcus aureus (Infections and infestations) | 1 (1)
Fungal Pneumonia (Infections and infestations) | 2 (2)
Infectious Diarrhea (Infections and infestations) | 6 (6)
Upper Respiratory Infection - Influenza A (Infections and infestations) | 5 (5)
Upper Respiratory Infection - SARS-CoV-2 (Infections and infestations) | 1 (1)
Upper Respiratory Infection - Coronavirus (Infections and infestations) | 2 (2)
Central Line Infection (Infections and infestations) | 4 (4)
Fungal Infection (Infections and infestations) | 1 (1)
Epstein Barr Virus Infection (Infections and infestations) | 9 (9)
Acute Graft-versus-Host Disease (Investigations) | 12 (12)
Platelet count decreased (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 3 (3)
Creatinine increased (Investigations) | 1 (1)
Chronic Graft-versus-Host Disease (Investigations) | 5 (5)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT02497404/Prot_SAP_000.pdf